CLINICAL TRIAL: NCT01755702
Title: A Study to Assess the Efficacy of Paracetamol Taken in Combination With Caffeine for the Treatment of Episodic Tension Type Headache
Brief Title: Paracetamol With Caffeine to Treat Episodic Tension Type Headache
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to unforeseen difficulties with subject recruitment. No safety issues were identified in the study with this new formulation.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A2260597
Record Dates: First submitted 2011-06-23; First posted 2012-12-24 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2014-11

CONDITIONS: Headache, Tension-Type
Keywords: caffeine; paracetamol; tension headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Arm 2 (Active Comparator): paracetamol marketed forumulation
  Interventions: Drug: Paracetamol marketed formulation
- Arm 3 (Active Comparator): ibuprofen marketed formulation
  Interventions: Drug: ibuprofen marketed formulation
- Arm 4 (Experimental): experimental paracetamol + caffeine formulation
  Interventions: Drug: Experimental paracetamol + caffeine formulation

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Arm 1
Drug: Experimental paracetamol + caffeine formulation — experimental paracetamol + caffeine formulation
  Arms: Arm 4
Drug: ibuprofen marketed formulation — ibuprofen marketed formulation
  Arms: Arm 3
Drug: Paracetamol marketed formulation — Paracetamol marketed formulation
  Arms: Arm 2

SUMMARY:
This study will compare a fast-absorbing paracetamol plus caffeine formula with placebo and an over-the-counter dose of paracetamol and ibuprofen to treat episodic tension headache.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of episodic tension-type headache consistent with all of the following:

  1. number of days with the condition is historically greater than or equal to two per month
  2. onset of condition was greater than or equal to 12 months from Visit 1
  3. age of onset was < 50 years
  4. severity of headaches is historically at least moderate
  5. duration of headaches is historically greater than or equal to four hours, if untreated
  6. number of headache episodes was greater than or equal to 4 and less than or equal to 10 during each of the three months immediately prior to Visit 1
  7. treatment of headache episodes with OTC analgesics has historically provided pain relief in less than or equal to 2 hours

Exclusion Criteria:

* Subject has chronic tension type headache, which is defined as headache on more than 15 days per month for 3 months.
* If a migraine sufferer,subject averages more than one episode per month, is incapable of differentiating between tension-type headaches and migraine headaches, and/or requires regular or prophylactic use of migraine medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Springfield Neurology Associates, Springfield, Massachusetts
  - MedVadis Research Corporation, Wellesley Hills, Massachusetts
  - Biomedical Research Alliance of New York LLC, Lake Success, New York
  - Elkind Headache Center, Mount Vernon, New York
  - International Research Service, Inc., Port Chester, New York
  - Jefferson Headache Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center study conducted at 7 centers.
Pre-assignment Details: 66 participants were randomized. Each participant was expected to complete 1, 2, or 3 periods depending on number of headache episodes, for example participants experiencing 2 episodes would take the first 2 treatments, but would not get the 3rd treatment. Such participants would be considered as completer, not a withdrawal.
Groups:
- Overall: In this cross-over study, participants were randomly-assigned to a blinded treatment sequence. Each participant was expected to complete 1, 2, or 3 periods depending on number of headache episodes.
  The following treatments were administered during the study.
  1. 1000/130mg paracetamol/caffeine (two 500/65mg caplets) plus placebo ibuprofen (two caplets) for a total of four caplets taken orally with approximately (approx.) 250 ml of water.
  2. 1000mg paracetamol (two 500mg caplets) plus placebo paracetamol/caffeine (two caplets) taken orally with approx. 250 ml of water.
  3. 400mg ibuprofen (two 200mg caplets) plus placebo paracetamol/caffeine (two caplets) for a total of four caplets taken orally with approx. 250 ml of water.
  4. placebo paracetamol/caffeine (two caplets) plus placebo ibuprofen (two caplets) for a total of four caplets taken orally with approx. 250 ml of water.
Period: Period I
Arm/Group | Overall
Started | 66
Received Paracetamol | 16
Received Placebo | 17
Received Ibuprofen | 16
Received Paracetamol/Caffeine | 17
Completed | 66
Not Completed | 0
Period: Wash Out Period I
Arm/Group | Overall
Started | 66
Completed | 63
Not Completed | 3
Not completed — Other Reason | 3
Period: Period II
Arm/Group | Overall
Started | 63
Received Ibuprofen | 11
Received Placebo | 15
Received Paracetamol/Caffeine | 20
Received Paracetamol | 17
Completed | 63
Not Completed | 0
Period: Washout Period II
Arm/Group | Overall
Started | 63
Completed | 58
Not Completed | 5
Not completed — Other Reason | 5
Period: Period III
Arm/Group | Overall
Started | 58
Received Paracetamol | 17
Received Placebo | 13
Received Paracetamol/Caffeine | 10
Received Ibuprofen | 18
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline measures.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.0 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Time to First Perceptible Headache Relief
Description: Time to first perceptible pain relief, calculated as time when partcipant selected 'a little' pain relief in the electronic pad minus the time of treatment. If this time was not available in the electronic pad then the earliest time corresponding to a pain relief score 1 or greater was recorded as time to 'a little' pain relief.
Time Frame: Baseline to 6 hours
Population: Intention to treat (ITT) population: All randomized participants who received at least one study medication and who had at least one post-baseline efficacy assessment.
Measure: Median (Full Range); unit: minutes
Groups:
- Paracetamol/Caffeine: Participants were administered with two paracetamol/ caffeine caplets (500/65 mg each) and two placebo caplets (matching ibuprofen) orally with approx. 250 mL of water.
- Ibuprofen: Participants were administered with two 200 mg Ibuprofen caplets and two placebo caplets (matching paracetamol/caffeine) orally with approx. 250 mL of water.
- Paracetamol: Participants were administered with two 500 mg paracetamol caplets and two placebo caplets (matching paracetamol/caffeine) orally with approx. 250 mL of water.
- Placebo: Participants were administered with four placebo caplets (two caplets matching paracetamol/caffeine and two caplets matching ibuprofen) orally with approx. 250 mL of water.
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
minutes | 30 [5 to 240] | 30 [8 to 120] | 30 [15 to 240] | 30 [12 to 240]
Statistical Analysis 1: Comparison: Paracetamol/Caffeine vs Placebo; Null hypothesis considered no difference between the treatments in comparison; Test type: Superiority or Other; p = 0.2840, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.83 to 1.90]
Statistical Analysis 2: Comparison: Paracetamol/Caffeine vs Paracetamol; Null hypothesis considered no difference between the treatments in comparison; Test type: Superiority or Other; p = 0.2008, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.86 to 2.01]
Statistical Analysis 3: Comparison: Paracetamol/Caffeine vs Ibuprofen; Null hypothesis considered no difference between the treatments in comparison; Test type: Superiority or Other; p = 0.4552, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.78 to 1.74]
Statistical Analysis 4: Comparison: Ibuprofen vs Paracetamol; Test type: Superiority or Other; p = 0.5579, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.75 to 1.71]
Statistical Analysis 5: Comparison: Ibuprofen vs Placebo; Null hypothesis considered no difference between the treatments in comparison; Test type: Superiority or Other; p = 0.7214, Cox Proportional Hazard Model; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.72 to 1.61]
Statistical Analysis 6: Comparison: Paracetamol vs Placebo; Null hypothesis considered no difference between the treatments in comparison; Test type: Superiority or Other; p = 0.8192, Cox Proportional Hazard Model; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.62 to 1.45]

2. Secondary Outcome: Headache Relief Scores
Description: Pain relief scores were measured on a scale from 0-4: 0- No pain relief; 1- Perceptible pain relief; 2- Meaningful pain relief; 3- A lot of relief and 4- Complete relief.
Time Frame: Baseline to 4 hours
Population: ITT population: All randomized participants who received at least one study medication and who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
Score on a scale
  15 minutes | 0.15 (0.427) | 0.08 (0.267) | 0.29 (0.622) | 0.08 (0.273)
  30 minutes | 1.09 (1.095) | 0.84 (0.754) | 0.81 (0.877) | 0.87 (0.951)
  45 minutes | 1.87 (0.894) | 1.61 (1.046) | 1.46 (0.969) | 1.70 (1.222)
  60 minutes | 2.79 (1.143) | 2.49 (1.023) | 2.05 (1.161) | 2.21 (1.277)
  90 minutes | 3.36 (0.903) | 3.16 (1.124) | 2.95 (1.280) | 2.95 (1.378)
  120 minutes | 3.50 (0.985) | 3.46 (1.141) | 3.35 (1.169) | 3.00 (1.414)
  240 minutes | 3.50 (1.012) | 3.75 (0.639) | 3.24 (1.179) | 3.55 (0.912)

3. Secondary Outcome: Total Pain Relief (TOTPAR)
Description: TOTPAR was calculated as sum of the products of pain relief score at time interval at 0-60 minutes, 60-90 minutes, 90-120 minutes and 120-240 minutes. Participants were asked to choose a number on a scale of 0 to 4, where, 0- No pain relief; 1- A little or perceptible pain relief; 2- Meaningful pain relief; 3- A lot of relief; 4- Complete relief. The mean PRS scores were calculated on the basis of participant's response based on the above score.
  It was calculated using the following formula.
  TOTPAR t = Σ(Rt x (time t - time t-1)), where Rt = pain relief score at time t; time t = time t in hours; time t-1 = time at previous time-point.
Time Frame: Baseline to 4 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
Score on a scale
  TOTPAR (0-60 minutes) | 1.57 (0.75) | 1.37 (0.64) | 1.14 (0.68) | 1.26 (0.82)
  TOTPAR (0-90 minutes) | 3.37 (1.08) | 2.96 (1.18) | 2.66 (1.20) | 2.79 (1.40)
  TOTPAR (0-120 minutes) | 5.08 (1.65) | 4.94 (1.63) | 4.62 (1.81) | 4.18 (1.97)
  TOTPAR (0-240 minutes) | 11.73 (3.22) | 12.08 (2.48) | 10.65 (3.74) | 11.19 (3.48)

4. Secondary Outcome: Sum of Pain Intensity Difference (SPID)
Description: Sum of pain intensity difference (SPID) at 60, 90, 120 and 240 minutes - calculated as the sum of headache intensity differences between the baseline pain intensity score and pain intensity score at each timepoint.
  Pain intensity was measured by numerical rating scale which is horizontal line with a scale from 0-10, where 0 represents no pain and 10 represents the worst possible pain.
  It was calculated using the following formula; SPID t = ΣPID x (time t - time t-1), where PID = PI (baseline) - PI t and PI = pain intensity.
Time Frame: Baseline to 4 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
Score on a scale
  SPID (0-60 minutes) | 1.49 (0.81) | 1.34 (0.64) | 1.15 (0.61) | 1.16 (0.72)
  SPID (0-90 minutes) | 3.06 (1.25) | 2.69 (1.13) | 2.48 (1.18) | 2.42 (1.20)
  SPID (0-120 minutes) | 4.42 (1.88) | 4.56 (1.73) | 4.32 (1.98) | 3.69 (1.70)
  SPID (0-240 minutes) | 9.43 (3.62) | 9.93 (3.28) | 8.69 (2.77) | 9.51 (3.29)

5. Secondary Outcome: Sum of TOTPAR and SPID (SPRID)
Description: Area under the time-response curve for change in headache intensity and headache relief (SPRID) at 60, 90, 120 and 240 minutes, was calculated as sum of TOTPAR and SPID:
  SPRIDt = TOTPARt + SPIDt
  TOTPAR was calculated as sum of the products of pain relief score. Participants were asked to choose a number on a scale of 0 to 4, where, 0- No pain relief; 1- A little or perceptible pain relief; 2- Meaningful pain relief; 3- A lot of relief; 4- Complete relief. The mean PRS scores were calculated on the basis of participant's response based on the above score.
  SPID was calculated as the sum of headache intensity differences between baseline and at each time point. It was measured by numerical rating scale which is horizontal line with a scale from 0-10, where 0 represents no pain and 10 represents the worst possible pain.
Time Frame: Baseline to 4 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
Score on a scale
  SPRID (0-60 minutes) | 3.05 (1.43) | 2.71 (1.19) | 2.28 (1.17) | 2.42 (1.47)
  SPRID (0-90 minutes) | 6.43 (2.17) | 5.66 (2.13) | 5.14 (2.26) | 5.22 (2.43)
  SPRID (0-120 minutes) | 9.50 (3.39) | 9.50 (3.08) | 8.94 (3.65) | 7.87 (3.34)
  SPRID (0-240 minutes) | 21.16 (6.18) | 22.00 (5.46) | 19.35 (5.72) | 20.70 (6.35)

6. Secondary Outcome: Time to Rescue Medication
Description: Time to rescue medication was evaluated.
Time Frame: Baseline to 6 hours post dose
Population: as for outcome 2
Measure: Median (Full Range); unit: minutes
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
minutes | 119.0 [119 to 119] | 150.0 [126 to 211] | 129.5 [129 to 130] | 62.0 [62 to 149]

7. Secondary Outcome: Number of Participants With Complete Headache Relief
Description: Number of headaches resolved at 1 and 2 hours before any rescue medication was calculated as number of participants with complete pain relief and headache severity of 'no headache' over total number of participants. These calculations were based on one headache per treatment per subject.
Time Frame: Baseline to 2 hours
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
Participants
  Headache resolved within 1 hour | 15 | 7 | 4 | 7
  Headache resolved within 2 hour | 29 | 30 | 25 | 24

8. Secondary Outcome: Headache Severity
Description: Headache severity (scores) at 15, 30, 45, 60, 90, 120, and 240 minutes were calculated as change (difference) from baseline of pain intensity at each time point.
  Pain intensity was measured by numerical rating scale which is a horizontal line with a scale from 0-10, where 0 represents no pain and 10 represents the worst possible pain.
Time Frame: Baseline to 4 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
Score on a scale
  15 minutes | 0.35 (0.802) | 0.20 (0.464) | 0.20 (0.406) | 0.18 (0.692)
  30 minutes | 1.03 (0.923) | 0.77 (0.649) | 0.78 (0.584) | 0.85 (0.779)
  45 minutes | 1.77 (0.986) | 1.61 (0.919) | 1.51 (0.823) | 1.38 (0.924)
  60 minutes | 2.50 (1.133) | 2.36 (1.013) | 2.00 (1.065) | 2.03 (1.102)
  90 minutes | 2.97 (1.063) | 2.76 (1.128) | 2.60 (1.172) | 2.57 (1.192)
  120 minutes | 2.94 (1.110) | 3.08 (1.100) | 2.94 (1.197) | 2.67 (1.238)
  240 minutes | 2.82 (0.958) | 3.05 (0.887) | 2.67 (0.856) | 3.00 (0.926)

9. Secondary Outcome: Patients Global Assessment in Response to Treatment
Description: Patients Global Assessment in Response to Treatment was assessed by a score in a scale from 0-4: 0- Poor; 1- Fair; 2- Good; 3- Very Good and 4- Excellent.
Time Frame: Baseline to 8 weeks
Population: as for outcome 2
Measure: Number; unit: Score on a scale
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Number analyzed (Participants) | 47 | 50 | 45 | 45
Score on a scale
  Score 0 (Very poor) | 1 | 1 | 1 | 2
  Score 1 (Poor) | 0 | 1 | 1 | 4
  Score 2 (Neutral) | 10 | 5 | 6 | 3
  Score 3 (Good) | 16 | 19 | 15 | 17
  Score 4 (Very Good) | 12 | 18 | 11 | 12

ADVERSE EVENTS:
Time Frame: All adverse events that occured in the time frame of start of the investigational product and until five days following last administration of the investigational product, were recorded.
Arm/Group | Paracetamol/Caffeine | Ibuprofen | Paracetamol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/50 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 2/47 | 4/50 | 0/45 | 3/45
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracetamol/Caffeine (N=47) | Ibuprofen (N=50) | Paracetamol (N=45) | Placebo (N=45)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar Fascilitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.